CLINICAL TRIAL: NCT05129553
Title: Béa Applicator and Béa Cervical Cap Usability Study
Brief Title: Béa Applicator and Béa Cervical Cap Safety and Usability Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: StepOne Fertility (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SOF63073301
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Safety and Usability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Use (Experimental): The participants will then be given the Béa Applicator and Béa Cervical Cap with accompanying instructions for single-use in a home use environment.
  Interventions: Device: Béa Applicator and Béa Cervical Cap Device

INTERVENTIONS:
Device: Béa Applicator and Béa Cervical Cap Device — Single-use of the investigational device

SUMMARY:
This is a Clinical Study Designed to Validate the Usability and Safety of the Over-the-counter (OTC) Béa Applicator and Béa Cervical Cap Device in a Home Use Environment.

DETAILED DESCRIPTION:
Female participants will undergo a baseline physical assessment performed by a physician at the study site. The participants will then be given the Béa Applicator and Béa Cervical Cap device with accompanying instructions and a semen collection pot. The participants will return home to use the device as per the Instruction for Use (IFU). The Béa Cervical Cap will remain in place for a minimum of 4 hours and a maximum of 6 hours. At the follow-up assessment, the investigator will investigate all primary objectives via a physical exam or via questioning the participant.

ELIGIBILITY:
Inclusion Criteria:

* People who are able to and for whom it is medically safe to conceive
* Heterosexual couples and individuals, of any race or ethnicity, who are sexually active
* 18 - 40 years of age
* Trying to conceive
* Signed Informed Consent
* Approximately nineteen per cent (19%) of participants will present with a retroverted uterus as found in the general female population.

Exclusion Criteria:

* Vaginal prolapse (female)
* Hysterectomy (female)
* Erectile dysfunction (male)
* Diagnosis and/or treatment of vaginitis or sexually transmitted infection (STI) within the last month
* Colposcopy with biopsy surgery within the last three (3) months (female)
* Treatment for dysplasia surgery within the previous three (3) months (female)
* Vaginal/cervical surgery within the last three (3) months (female)
* Current pregnancy (female)
* Unable to read and understand English, as assessed by REALM
* Presence of noticeable lesions, open sores, viral warts, and any other genital abnormalities (female & male)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Correctly place semen in the device | 0.5 hrs
  Participants indicate an ability to collect and transfer semen into the device in the intended use environment (at-home).
Correctly inserting the device into the vagina | 1 hrs
  Participants indicate an ability to insert the device into the vagina, in the intended use environment (at-home).
Correctly positioning of the device over the cervical os | 4-6 hrs
  A clinical examination by a physician to confirm the device is positioned over the cervical os.
Correctly withdraw the device from the vagina | 4-6 hrs
  Participants indicate an ability to withdraw the device from the vagina with the use of the removal string.
The device causes trauma or harm | 4-6 hrs
  After the device is removed from the vagina, a physician assessment via a speculum examination to determine if the device caused trauma or harm to the vaginal epithelium or cervix.
Presence of semen in the cap | 4-6 hrs
  After the device is removed from the vagina, a physician assesses the presence of semen remaining in the cervical cap.
Correctly dispose of the used device after use | 4-6 hrs
  Participants indicate an ability to dispose of the device after use.
Correctly avoid sexual activity while the device is in place | 4-6 hrs
  Participants indicate an ability to avoid sexual activity while the device is on the cervical os.

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared with researchers outside the study.